CLINICAL TRIAL: NCT00567580
Title: A Phase III Trial of Short Term Androgen Deprivation With Pelvic Lymph Node or Prostate Bed Only Radiotherapy (SPPORT) in Prostate Cancer Patients With a Rising PSA After Radical Prostatectomy
Brief Title: Prostate Radiation Therapy or Short-Term Androgen Deprivation Therapy and Pelvic Lymph Node Radiation Therapy With or Without Prostate Radiation Therapy in Treating Patients With a Rising Prostate Specific Antigen (PSA) After Surgery for Prostate Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); Cancer and Leukemia Group B (Network); NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RTOG-0534; CDR0000577574; NCI-2009-00733 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCT01312974 (obsolete NCT alias)
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Results first posted 2021-03-02 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-05

CONDITIONS: Prostate Cancer
Keywords: stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated; Flutamide; bicalutamide; Gonadotropin-Releasing Hormone; Leuprolide; Goserelin; Buserelin; Triptorelin Pamoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PBRT Alone (Active Comparator): Prostate bed radiotherapy (PBRT) begins within 6 weeks (+/- 2 weeks) after registration.
  Interventions: Radiation: PBRT
- PBRT + STAD (Experimental): Prostate bed radiotherapy (PBRT) and short term androgen deprivation therapy (STAD) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STAD starts first, 2 months (+/- 2 weeks) before radiotherapy (RT), and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
  Interventions: Radiation: PBRT; Drug: AA; Drug: LHRH agonist
- PLNRT + PBRT + STADT (Experimental): Pelvic lymph node radiotherapy (PLNRT), prostate bed radiotherapy (PBRT), and short term androgen deprivation therapy (STAD) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STAD starts first, 2 months (+/- 2 weeks) before RT, and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
  Interventions: Radiation: PBRT; Radiation: PLNRT; Drug: AA; Drug: LHRH agonist

INTERVENTIONS:
Radiation: PBRT — 1.8 Gy per fraction once daily, 5 days a week totaling 64.8-70.2 Gy. 3D-CRT or IMRT required.
  Other Names: Prostate bed radiotherapy; Three-Dimensional Conformal Radiation Therapy (3D-CRT); Intensity modulated RT (IMRT)
Radiation: PLNRT — 1.8 Gy per fraction once daily, 5 days a week, totaling 45 Gy. 3D-CRT or IMRT required.
  Other Names: Pelvic lymph node radiotherapy
  Arms: PLNRT + PBRT + STADT
Drug: AA — Antiandrogen (AA) therapy can be either 250 mg flutamide by mouth three times a day or 50 mg bicalutamide by mouth once a day.
  Other Names: flutamide; bicalutamide
  Arms: PBRT + STAD; PLNRT + PBRT + STADT
Drug: LHRH agonist — Luteinizing hormone-releasing hormone (LHRH) agonist can be any analog approved by the FDA (or by Health Canada for Canadian institutions) and may be given in any possible combination such that the total LHRH treatment time is 4-6 months. LHRH analogs are administered with a variety of techniques, including subcutaneous insertion of a solid plug in the abdominal wall, intramuscular injection, and subcutaneous injection.
  Other Names: leuprolide; goserelin; buserelin; triptorelin
  Arms: PBRT + STAD; PLNRT + PBRT + STADT

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as flutamide, bicalutamide, and luteinizing hormone-releasing hormone agonist, may lessen the amount of androgens made by the body. It is not yet known which regimen of radiation therapy with or without androgen-deprivation therapy is more effective for prostate cancer.

PURPOSE: This randomized phase III trial is studying prostate radiation therapy to see how well it works compared with short-term androgen deprivation therapy given together with pelvic lymph node radiation therapy with or without prostate radiation therapy in treating patients with a rising PSA after surgery for prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine whether the addition of short-term androgen deprivation (STAD) to prostate bed radiotherapy (PBRT) improves freedom from progression (FFP) (i.e., maintenance of a prostate-specific antigen [PSA] less than the nadir+2 ng/mL, absence of clinical failure, and absence of death from any cause) for 5 years, over that of PBRT alone in men treated with salvage radiotherapy after radical prostatectomy.
* To determine whether STAD, pelvic lymph node radiotherapy (PLNRT), and PBRT improves FFP over that of STAD+PBRT and PBRT alone in men treated with salvage radiotherapy after radical prostatectomy.

Secondary

* To compare secondary biochemical failure, the development of hormone-refractory disease , distant metastasis, cause-specific mortality, and overall mortality at five years.
* To compare acute and late morbidity based on Common Toxicity Criteria for Adverse Effects (CTCAE), v. 3.0.
* To measure the expression of cell kinetic, apoptotic pathway, and angiogenesis-related genes in archival diagnostic tissue to better define the risk of FFP, distant failure, cause-specific mortality, and overall mortality after salvage radiotherapy for prostate cancer, independently of conventional clinical parameters now used.
* To quantify blood product-based proteomic and genomic (single nucleotide polymorphisms) patterns and urine-based genomic patterns before and at different times after treatment to better define the risk of FFP, distant failure, cause-specific mortality, and overall mortality after salvage radiotherapy for prostate cancer, independently of conventional clinical parameters now used.
* To assess the degree, duration, and significant differences of disease-specific health-related quality of life (HRQOL) decrements among treatment arms.
* To assess whether mood is improved and depression is decreased with the more aggressive therapy if it improves FFP.
* To collect paraffin-embedded tissue blocks, serum, plasma, urine, and buffy coat cells for future translational research analyses.

Tertiary

* To assess whether an incremental gain in FFP and survival with more aggressive therapy outweighs decrements in the primary generic domains of HRQOL (i.e., mobility, self care, usual activities, pain/discomfort, and anxiety/depression).
* To evaluate the cost-utility of the treatment arm demonstrating the most significant benefit (in terms of the primary outcome) in comparison with other widely accepted cancer and non-cancer therapies.
* To assess associations between serum levels of beta-amyloid and measures of cognition and mood and depression.
* An exploratory aim is to assess the relationship(s) between the American Urological Association Symptom Index (AUA SI) and urinary morbidity using the CTCAE v. 3.0 grading system.

OUTLINE: Patients are stratified according to seminal vesicle involvement (yes vs no), prostatectomy Gleason score (≤ 7 vs 8-9), pre-radiotherapy PSA (≥ 0.1 and ≤ 1.0 ng/mL vs > 1.0 and < 2.0 ng/mL), and pathology stage (pT2 and margin negative vs all others). Patients are randomized to 1 of 3 treatment arms.

Follow-up occurs 3, 6, and 12 months after the completion of radiation therapy, then every 6 months for 6 years, and then annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Adenocarcinoma of the prostate treated primarily with radical prostatectomy, pathologically proven to be lymph node negative by pelvic lymphadenectomy (N0) or lymph node status pathologically unknown (undissected pelvic lymph nodes [Nx]), i.e. lymph node dissection is not required;

   • Any type of radical prostatectomy will be permitted, including retropubic, perineal, laparoscopic or robotically assisted. There is no time limit for the date of radical prostatectomy.
2. A post-radical prostatectomy entry prostate-specific antigen (PSA) of ≥ 0.1 and < 2.0 ng/mL at least 6 weeks (45 days) after prostatectomy and within 30 days of registration;
3. One of the following pathologic classifications:

   * T3N0/Nx disease with or without a positive prostatectomy surgical margin; or
   * T2N0/Nx disease with or without a positive prostatectomy surgical margin;
4. Prostatectomy Gleason score of 9 or less;
5. Zubrod Performance Status of 0-1;
6. Age ≥ 18;
7. No distant metastases, based upon the following minimum diagnostic workup:

   * History/physical examination (including digital rectal exam) within 8 weeks (60 days) prior to registration;
   * A computerized tomography (CT) scan of the pelvis (with contrast if renal function is acceptable; a noncontrast CT is permitted if the patient is not a candidate for contrast) or magnetic resonance imaging (MRI) of the pelvis within 120 days prior to registration;
   * Bone scan within 120 days prior to registration; if the bone scan is suspicious, a plain x-ray and/or MRI must be obtained to rule out metastasis.
8. Adequate bone marrow function, within 90 days prior to registration, defined as follows:

   * Platelets ≥ 100,000 cells/mm^3 based upon compete blood count (CBC);
   * Hemoglobin ≥ 10.0 g/dl based upon CBC (Note: The use of transfusion or other intervention to achieve Hgb ≥ 10.0 g/dl is recommended).
9. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) < 2 x the upper limit of normal within 90 days prior to registration;
10. Serum total testosterone must be ≥ 40% of the lower limit of normal (LLN) of the assay used (testosterone ÷ LLN must be ≥ 0.40) within 90 days prior to registration (Note: Patients who have had a unilateral orchiectomy are eligible as long as this requirement is met);
11. Patients must sign a study-specific informed consent prior to study entry.

Exclusion Criteria:

1. A palpable prostatic fossa abnormality/mass suggestive of recurrence, unless shown by biopsy under ultrasound guidance not to contain cancer;
2. N1 patients are ineligible, as are those with pelvic lymph node enlargement ≥ 1.5 cm in greatest dimension by CT scan or MRI of the pelvis, unless the enlarged lymph node is sampled and is negative;
3. Androgen deprivation therapy started prior to prostatectomy for > 6 months (180 days) duration. Note: The use of finasteride or dutasteride (±tamsulosin) for longer periods prior to prostatectomy is acceptable;
4. Androgen deprivation therapy started after prostatectomy and prior to registration (Note: The use of finasteride or dutasteride (±tamsulosin) after prostatectomy is not acceptable - must be stopped within 3 months after prostatectomy. Androgen deprivation therapy must be stopped within 3 months after prostatectomy);
5. Neoadjuvant chemotherapy before or after prostatectomy;
6. Prior chemotherapy for any other disease site if given within 5 years prior to registration;
7. Prior cryosurgery or brachytherapy of the prostate; prostatectomy should be the primary treatment and not a salvage procedure;
8. Prior pelvic radiotherapy;
9. Prior invasive malignancy (except non-melanomatous skin cancer) or superficial bladder cancer unless disease free for a minimum of 5 years [for example, carcinoma in situ of the oral cavity is permissible];
10. Severe, active co-morbidity, defined as follows:

    * History of inflammatory bowel disease;
    * History of hepatitis B or C; Blood tests are not required to determine if the patient has had hepatitis B or C, unless the patient reports a history of hepatitis.
    * Unstable angina and/or congestive heart failure requiring hospitalization within the last 6 months;
    * Transmural myocardial infarction within the last 6 months;
    * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration;
    * Chronic Obstructive Pulmonary Disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration;
    * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; AST or ALT are required; note, however, that laboratory tests for coagulation parameters are not required for entry into this protocol.
    * Acquired Immune Deficiency Syndrome (AIDS) based upon current Centers for Disease Control and Prevention (CDC) definition; Note, however, that human immunodeficiency viruses (HIV) testing is not required for entry into this protocol. The need to exclude patients with acquired immunodeficiency syndrome (AIDS) from this protocol is necessary because the treatments involved in this protocol may result in increased toxicity and immunosuppression.
11. Prior allergic reaction to the study drug(s) involved in this protocol.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1792 (Actual)
Dates: Start 2008-02; Primary Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan Pollack, MD, PhD, Principal Investigator — University of Miami
Locations (460):
- United States (444):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Fairbanks Cancer Treatment Center at Fairbanks Memorial Hospital, Fairbanks, Alaska
  - Arizona Center for Cancer Care - Peoria, Peoria, Arizona
  - Arizona Oncology Services Foundation, Phoenix, Arizona
  - Arizona Oncology - Tucson, Tucson, Arizona
  - Auburn Radiation Oncology, Auburn, California
  - Peninsula Medical Center, Burlingame, California
  - Radiation Oncology Centers - Cameron Park, Cameron Park, California
  - Mercy Cancer Center at Mercy San Juan Medical Center, Carmichael, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Valley Medical Oncology Consultants - Castro Valley, Castro Valley, California
  - Enloe Cancer Center at Enloe Medical Center, Chico, California
  - Valley Medical Oncology, Fremont, California
  - Washington Township Hospital, Fremont, California
  - California Cancer Center - Woodward Park Office, Fresno, California
  - Cancer Care Associates, Fresno, California
  - Rebecca and John Moores UCSD Cancer Center, La Jolla, California
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - Samuel Oschin Comprehensive Cancer Institute at Cedars-Sinai Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center and Hospital, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Providence Holy Cross Cancer Center, Mission Hills, California
  - Memorial Medical Center, Modesto, California
  - El Camino Hospital Cancer Center, Mountain View, California
  - Sutter Health - Western Division Cancer Research Group, Novato, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons, Incorporated, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee, Incorporated, Oakland, California
  - St. Joseph Hospital Regional Cancer Center - Orange, Orange, California
  - Feather River Hospital Cancer Center, Paradise, California
  - Radiation Oncology Center - Roseville, Roseville, California
  - Radiological Associates of Sacramento Medical Group, Incorporated, Sacramento, California
  - University of California Davis Cancer Center, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - California Pacific Medical Center - California Campus, San Francisco, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Saint Helena Hospital, St. Helena, California
  - Solano Radiation Oncology Center, Vacaville, California
  - Sutter Solano Medical Center, Vallejo, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Middlesex Hospital Cancer Center, Middletown, Connecticut
  - George Bray Cancer Center at the Hospital of Central Connecticut - New Britain Campus, New Britain, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - CCOP - Christiana Care Health Services, Newark, Delaware
  - Washington Cancer Institute at Washington Hospital Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Integrated Community Oncology Network at Southside Cancer Center, Jacksonville, Florida
  - Baptist Medical Center South, Jacksonville, Florida
  - Integrated Community Oncology Network, Jacksonville Beach, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Integrated Community Oncology Network - Orange Park, Orange Park, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - Florida Cancer Center - Palatka, Palatka, Florida
  - Flagler Cancer Center, Saint Augustine, Florida
  - Veterans Affairs Medical Center - Tampa, Tampa, Florida
  - Emory Crawford Long Hospital, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - John B. Amos Cancer Center, Columbus, Georgia
  - Northside Hospital-Forsyth, Cumming, Georgia
  - Piedmont Fayette Hospital, Fayetteville, Georgia
  - Nancy N. and J. C. Lewis Cancer and Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - Hawaii Medical Center - East, Honolulu, Hawaii
  - Pacific Cancer Institute - Maui, Wailuku, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - Saint Alphonsus Cancer Care Center at Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Creticos Cancer Center at Advocate Illinois Masonic Medical Center, Chicago, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Leonard C. Ferguson Cancer Center, Freeport, Illinois
  - Ingalls Cancer Care Center at Ingalls Memorial Hospital, Harvey, Illinois
  - Veterans Affairs Medical Center - Hines, Hines, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Trinity Cancer Center at Trinity Medical Center - 7th Street Campus, Moline, Illinois
  - Cancer Institute at St. John's Hospital, Springfield, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Radiation Oncology Associates Southwest, Fort Wayne, Indiana
  - Parkview Regional Cancer Center at Parkview Health, Fort Wayne, Indiana
  - Center for Cancer Care at Goshen General Hospital, Goshen, Indiana
  - Howard Community Hospital, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Saint Joseph Regional Medical Center, Mishawaka, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Norton Suburban Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - Mary Bird Perkins Cancer Center - Baton Rouge, Baton Rouge, Louisiana
  - MBCCOP - LSU Health Sciences Center, New Orleans, Louisiana
  - Medical Center of Louisiana - New Orleans, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center Cancer Center, Baltimore, Maryland
  - St. Agnes Hospital Cancer Center, Baltimore, Maryland
  - Central Maryland Oncology Center, Columbia, Maryland
  - Tate Cancer Center at Baltimore Washington Medical Center, Glen Burnie, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana-Farber Cancer Institute, Boston, Massachusetts
  - Boston University Cancer Research Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Hudner Oncology Center at Saint Anne's Hospital - Fall River, Fall River, Massachusetts
  - Cape Cod Hospital, Hyannis, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - Saint Joseph Mercy Cancer Center, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Henry Ford Macomb Hospital, Clinton Township, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - McLaren Cancer Institute, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Foote Memorial Hospital, Jackson, Michigan
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - St. Mary Mercy Hospital, Livonia, Michigan
  - St. Joseph Mercy Oakland, Pontiac, Michigan
  - Mercy Regional Cancer Center at Mercy Hospital, Port Huron, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Seton Cancer Institute at Saint Mary's - Saginaw, Saginaw, Michigan
  - Lakeland Regional Cancer Care Center - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - MeritCare Bemidji, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - St. Luke's Hospital Cancer Care Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Immanuel St. Joseph's, Mankato, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Willmar Cancer Center at Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology - Woodbury, Woodbury, Minnesota
  - Regional Cancer Center at Singing River Hospital, Pascagoula, Mississippi
  - Cancer Institute of Cape Girardeau, LLC, Cape Girardeau, Missouri
  - Siteman Cancer Center at Barnes-Jewish St. Peters Hospital - St. Peters, City of Saint Peters, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital - Saint Louis, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Sletten Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - Saint Elizabeth Cancer Institute at Saint Elizabeth Regional Medical Center, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Methodist Estabrook Cancer Center, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Lakeside Hospital, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Center for Cancer Care at Exeter Hospital, Exeter, New Hampshire
  - Kingsbury Center for Cancer Care at Cheshire Medical Center, Keene, New Hampshire
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Memorial Sloan-Kettering Cancer Center - Basking Ridge, Basking Ridge, New Jersey
  - AtlantiCare Cancer Care Institute at AtlantiCare Regional Medical Center - Mainland Campus, Galloway, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Capital Health Regional Cancer Center, Pennington, New Jersey
  - Valley Hospital - Ridgewood, Ridgewood, New Jersey
  - Somerset Medical Center, Somerville, New Jersey
  - Frederick R. and Betty M. Smith Cancer Treatment Center, Sparta, New Jersey
  - Franklin & Edith Scarpa Regional Cancer Center at South Jersey Healthcare, Vineland, New Jersey
  - Cancer Institute of New Jersey at Cooper - Voorhees, Voorhees Township, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - University of New Mexico Cancer Center - South, Las Cruces, New Mexico
  - New York Oncology Hematology, PC at Albany Regional Cancer Care, Albany, New York
  - New York Methodist Hospital, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Sands Cancer Center, Canandaigua, New York
  - Memorial Sloan-Kettering Cancer Center, Commack, New York
  - Stich Radiation Center at NewYork-Presbyterian Hospital/Weill Cornell Medical Center, New York, New York
  - St. Luke's - Roosevelt Hospital Center - St.Luke's Division, New York, New York
  - Dyson Center for Cancer Care at Vassar Brothers Medical Center, Poughkeepsie, New York
  - Hudson Valley Oncology Associates, Poughkeepsie, New York
  - Highland Hospital of Rochester, Rochester, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - University Radiation Oncology at Parkridge Hospital, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan-Kettering Cancer Center - Rockville Centre, Rockville Centre, New York
  - Memorial Sloan-Kettering Cancer Center at Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - Randolph Hospital, Asheboro, North Carolina
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Moses Cone Regional Cancer Center at Wesley Long Community Hospital, Greensboro, North Carolina
  - Coleman Radiation Oncology Center at Carter General Hospital, Morehead City, North Carolina
  - CarolinaEast Cancer Care, New Bern, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Rex Cancer Center at Rex Hospital, Raleigh, North Carolina
  - Annie Penn Cancer Center, Reidsville, North Carolina
  - South Atlantic Radiation Oncology, LLC, Supply, North Carolina
  - Coastal Carolina Radiation Oncology Center, Wilmington, North Carolina
  - Zimmer Cancer Center at New Hanover Regional Medical Center, Wilmington, North Carolina
  - MeritCare Broadway, Fargo, North Dakota
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Roger Maris Cancer Center at MeritCare Hospital, Fargo, North Dakota
  - Altru Cancer Center at Altru Hospital, Grand Forks, North Dakota
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Summa Center for Cancer Care at Akron City Hospital, Akron, Ohio
  - Barberton Citizens Hospital, Barberton, Ohio
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Cancer Center at Fairview Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Arthur G. James Cancer Hospital and Richard J. Solove Research Institute at Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Medical Center Cancer Care, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Community Cancer Center, Elyria, Ohio
  - Hematology Oncology Center, Elyria, Ohio
  - Cleveland Clinic Cancer Center, Independence, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Hillcrest Cancer Center at Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake/University Ireland Cancer Center, Mentor, Ohio
  - Southwest General Health Center, Middleburg Heights, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - UHHS Chagrin Highlands Medical Center, Orange, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Parma Community General Hospital, Parma, Ohio
  - Southern Ohio Medical Center Cancer Center, Portsmouth, Ohio
  - Cancer Care Center, Incorporated, Salem, Ohio
  - North Coast Cancer Care, Incorporated, Sandusky, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Tony Teramana Cancer Center, Steubenville, Ohio
  - Cleveland Clinic Foundation - Strongsville, Strongsville, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - St. Anne Mercy Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - Mount Carmel St. Ann's Cancer Center, Westerville, Ohio
  - UHHS Westlake Medical Center, Westlake, Ohio
  - Cancer Treatment Center, Wooster, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at St. Francis Hospital, Tulsa, Oklahoma
  - Willamette Valley Cancer Center - Eugene, Eugene, Oregon
  - Three Rivers Community Hospital, Grants Pass, Oregon
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Dubs Cancer Center at Rogue Valley Medical Center, Medford, Oregon
  - Providence Cancer Center at PMCC, Medford, Oregon
  - Legacy Good Samaritan Hospital & Comprehensive Cancer Center, Portland, Oregon
  - Salem Hospital Regional Cancer Care Services, Salem, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rosenfeld Cancer Center at Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Cancer Center at Beaver Medical Center, Beaver, Pennsylvania
  - St. Luke's Cancer Network at St. Luke's Hospital, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - UPMC Cancer Center at Jefferson Regional Medical Center, Clairton, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Northeast Radiation Oncology Center, Dunmore, Pennsylvania
  - Adams Cancer Center, Gettysburg, Pennsylvania
  - UPMC Cancer Center - Arnold Palmer Pavilion, Greensburg, Pennsylvania
  - Penn State Hershey Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - UPMC Cancer Center at the John P. Murtha Pavilion, Johnstown, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - St. Mary Regional Cancer Center, Langhorne, Pennsylvania
  - UPMC Cancer Center at UPMC McKeesport, McKeesport, Pennsylvania
  - Upper Delaware Valley Cancer Center, Milford, Pennsylvania
  - Intercommunity Cancer Center, Monroeville, Pennsylvania
  - UPMC - Moon, Moon Township, Pennsylvania
  - Alle-Kiski Medical Center, Natrona Heights, Pennsylvania
  - UPMC Cancer Center - Natrona Heights, Natrona Heights, Pennsylvania
  - Jameson Memorial Hospital - North Campus, New Castle, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Kimmel Cancer Center at Thomas Jefferson University - Philadelphia, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - Albert Einstein Cancer Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC - Shadyside, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Presbyterian, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC St. Margaret, Pittsburgh, Pennsylvania
  - UPMC Cancer Center at UPMC Passavant, Pittsburgh, Pennsylvania
  - UPMC Cancer Center - Upper St. Clair, Pittsburgh, Pennsylvania
  - St. Joseph Medical Center, Reading, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Washington Hospital Cancer Center, Washington, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - Main Line Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - York Cancer Center at Apple Hill Medical Center, York, Pennsylvania
  - AnMed Cancer Center, Anderson, South Carolina
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Cancer Centers of the Carolinas - Faris Road, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Grove Commons, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Eastside, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Cancer Centers of the Carolinas - Greer Medical Oncology, Greer, South Carolina
  - Cancer Centers of the Carolinas - Greer Radiation Oncology, Greer, South Carolina
  - Hilton Head Radiation Oncology Center, Hilton Head Island, South Carolina
  - Cancer Centers of the Carolinas - Seneca, Seneca, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Cancer Centers of the Carolinas - Spartanburg, Spartanburg, South Carolina
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - West Tennessee Cancer Center at Jackson-Madison County General Hospital, Jackson, Tennessee
  - Texas Oncology, PA at Harris Center HEB, Bedford, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Texas Oncology, PA at Texas Cancer Center - Denton South, Denton, Texas
  - Klabzuba Cancer Center at Harris Methodist Fort Worth Hospital, Fort Worth, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Memorial Hermann Hospital - Memorial City, Houston, Texas
  - Texas Oncology, PA at Lake Vista Cancer Center, Lewisville, Texas
  - Longview Cancer Center, Longview, Texas
  - Cancer Care Centers of South Texas - Northeast, San Antonio, Texas
  - Texas Oncology, PA at Texas Cancer Center - Sherman, Sherman, Texas
  - Texas Oncology, PA at Texas Oncology Cancer Center Sugar Land, Sugar Land, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Texas Oncology, PA - Wichita Falls, Wichita Falls, Texas
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - Val and Ann Browning Cancer Center at McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Norris Cotton Cancer Center - North, Saint Johnsbury, Vermont
  - INOVA Alexandria Hospital, Alexandria, Virginia
  - Martha Jefferson Hospital Cancer Care Center, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Sentara Cancer Institute at Sentara Norfolk General Hospital, Norfolk, Virginia
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Veterans Affairs Medical Center - Richmond, Richmond, Virginia
  - Coastal Cancer Center at Sentara Virginia Beach General Hospital, Virginia Beach, Virginia
  - St. Joseph Cancer Center, Bellingham, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Franciscan Cancer Center at St. Joseph Medical Center, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - Legacy Salmon Creek Medical Center, Vancouver, Washington
  - North Star Lodge Cancer Center at Yakima Valley Memorial Hospital, Yakima, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Langlade Memorial Hospital, Antigo, Wisconsin
  - Fox Valley Hematology and Oncology - East Grant Street, Appleton, Wisconsin
  - Theda Care Cancer Institute, Appleton, Wisconsin
  - Beloit Memorial Hospital, Beloit, Wisconsin
  - Central Wisconsin Cancer Program at Agnesian HealthCare, Fond du Lac, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Franciscan Skemp Healthcare - La Crosse Campus, La Crosse, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Community Memorial Hospital Cancer Care Center, Menomonee Falls, Wisconsin
  - Columbia Saint Mary's Hospital - Ozaukee, Mequon, Wisconsin
  - Columbia-Saint Mary's Water Tower Medical Commons, Milwaukee, Wisconsin
  - Vince Lombardi Cancer Clinic at Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Veterans Affairs Medical Center - Milwaukee, Milwaukee, Wisconsin
  - D.N. Greenwald Center, Mukwonago, Wisconsin
  - Regional Cancer Center at Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - All Saints Cancer Center at Wheaton Franciscan Healthcare, Racine, Wisconsin
  - Door County Cancer Center at Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Aurora Medical Center, Summit, Wisconsin
  - Waukesha Memorial Hospital Regional Cancer Center, Waukesha, Wisconsin
  - University of Wisconcin Cancer Center at Aspirus Wausau Hospital, Wausau, Wisconsin
  - West Allis Memorial Hospital, West Allis, Wisconsin
  - Riverview UW Cancer Center at Riverview Hospital, Wisconsin Rapids, Wisconsin
  - Rocky Mountain Oncology, Casper, Wyoming
- Canada (13):
  - Tom Baker Cancer Centre - Calgary, Calgary, Alberta
  - Cross Cancer Institute at University of Alberta, Edmonton, Alberta
  - Saint John Regional Hospital, Saint John, New Brunswick
  - Doctor H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - Margaret and Charles Juravinski Cancer Centre, Hamilton, Ontario
  - London Regional Cancer Program at London Health Sciences Centre, London, Ontario
  - Cancer Care Program at Thunder Bay Regional Health Sciences, Thunder Bay, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
  - CHUS-Hopital Fleurimont, Sherbrooke, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
- Pamela Youde Nethersole Eastern Hospital, Hong Kong, China
- Israel (2):
  - Rabin Medical Center - Beilinson Campus, Petah Tikva
  - Tel-Aviv Sourasky Medical Center, Tel Aviv

REFERENCES:
- [Derived] Pollack A, Karrison TG, Balogh AG, Gomella LG, Low DA, Bruner DW, Wefel JS, Martin AG, Michalski JM, Angyalfi SJ, Lukka H, Faria SL, Rodrigues GB, Beauchemin MC, Lee RJ, Seaward SA, Allen AM, Monitto DC, Seiferheld W, Sartor O, Feng F, Sandler HM. The addition of androgen deprivation therapy and pelvic lymph node treatment to prostate bed salvage radiotherapy (NRG Oncology/RTOG 0534 SPPORT): an international, multicentre, randomised phase 3 trial. Lancet. 2022 May 14;399(10338):1886-1901. doi: 10.1016/S0140-6736(21)01790-6. PMID 35569466
- Available data/document: Individual Participant Data Set: NCT00567580 — https://nctn-data-archive.nci.nih.gov/ — Select individual patient-level data from this trial can be requested from the NCTN/NCORP Data Archive

RESULTS

PARTICIPANT FLOW:
Groups:
- PLNRT + PBRT + STAD: Pelvic lymph node radiotherapy (PLNRT), prostate bed radiotherapy (PBRT), and short term androgen deprivation therapy (STAD) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STAD starts first, 2 months (+/- 2 weeks) before RT, and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
Period: Overall Study
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Started | 592 | 602 | 598
Eligible | 564 | 578 | 574
Eligible, Started Study Treatment, and Have Adverse Event Data | 547 | 563 | 563
Completed (Participants contributing data to analysis are considered to have completed the study.) | 564 | 578 | 574
Not Completed | 28 | 24 | 24
Not completed — Protocol Violation | 28 | 24 | 24

BASELINE CHARACTERISTICS:
Population: Eligible participants
Groups:
- Total: Total of all reporting groups
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD | Total
Number analyzed (Participants) | 564 | 578 | 574 | 1716
Age, Continuous [Median (Full Range); unit: years] | 64 [42 to 84] | 64 [39 to 80] | 64 [44 to 80] | 64 [39 to 84]
Age, Customized [Count of Participants; unit: Participants]
  Age (years): <=49 | 19 | 15 | 8 | 42
  Age (years): 50-59 | 118 | 137 | 138 | 393
  Age (years): 60-69 | 307 | 299 | 307 | 913
  Age (years): >=70 | 120 | 127 | 121 | 368
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 564 | 578 | 574 | 1716
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 23 | 30 | 74
  Not Hispanic or Latino | 511 | 527 | 517 | 1555
  Unknown or Not Reported | 32 | 28 | 27 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 5 | 5
  Asian | 3 | 6 | 8 | 17
  Native Hawaiian or Other Pacific Islander | 1 | 4 | 0 | 5
  Black or African American | 74 | 69 | 77 | 220
  White | 464 | 482 | 474 | 1420
  More than one race | 3 | 0 | 0 | 3
  Unknown or Not Reported | 19 | 17 | 10 | 46
Zubrod Performance Status [Count of Participants; unit: Participants] — 0 = Asymptomatic; 1 = Symptomatic but completely ambulatory; 2 = Symptomatic, <50% in bed during the day; 3 = Symptomatic, >50% in bed, but not bedbound; 4 = Bedbound; 5 = Death
  Participants
    0 | 522 | 539 | 540 | 1601
    1 | 42 | 39 | 34 | 115
Pathologic Seminal Vesicle Involvement [Count of Participants; unit: Participants]
  No | 482 | 494 | 488 | 1464
  Yes | 82 | 84 | 86 | 252
Prostatectomy Tumor Stage [Count of Participants; unit: Participants] — Tumor stage per the American Joint Committee on Cancer (AJCC) 6th ed. refers to the size and/or extent of the main tumor. The higher the number after the T, the larger the tumor or the more it has grown into nearby tissues. T's may be further divided to provide more detail, such as T3a and T3b.
  Participants
    pT2 | 292 | 317 | 304 | 913
    pT3 Extraprostatic extension NOS | 13 | 15 | 18 | 46
    pT3a Extraprostatic extension | 177 | 162 | 166 | 505
    pT3b Seminal vesicle invasion | 82 | 84 | 86 | 252
Gleason Score [Count of Participants; unit: Participants] — Gleason score describes prostate cancer based on how abnormal the cancer cells in a biopsy sample look under a microscope. Cells are scored 1-5 with 1 indicating "low-grade" looking similar to normal cells and 5 indicating "high-grade" barely resembling normal cells due to mutation. A pathologist assigns a Gleason grade to the first and second most predominant patterns in the biopsy. The two grades are added together to calculate the Gleason score (between 2 and 10). Cancers with lower scores tend to be less aggressive, while cancers with higher scores end to be more aggressive.
  Participants
    4 | 0 | 1 | 1 | 2
    5 | 3 | 1 | 5 | 9
    6 | 80 | 85 | 89 | 254
    7: 3+4 | 226 | 240 | 221 | 687
    7:4+3 | 153 | 148 | 156 | 457
    7: primary/secondary not indicated | 9 | 5 | 3 | 17
    8 | 57 | 60 | 57 | 174
    9 | 36 | 38 | 42 | 116
Prostatectomy Margins [Count of Participants; unit: Participants]
  Positive | 288 | 289 | 284 | 861
  Negative | 267 | 284 | 287 | 838
  Unknown | 9 | 5 | 3 | 17
Pelvic Lymphadenectomy [Count of Participants; unit: Participants]
  No | 189 | 207 | 209 | 605
  Yes | 375 | 371 | 365 | 1111
Number of Lymph Nodes Examined [Median (Full Range); unit: lymph nodes] — Population: Eligible with lymphadenectomy details
  lymph nodes
    number analyzed (Participants) | 349 | 336 | 336 | 1021
    (all) | 5 [0 to 34] | 6 [1 to 54] | 5 [1 to 32] | 6 [0 to 54]
Pre-RT Entry PSA [Median (Full Range); unit: ng/ml] — Prostate-specific antigen (PSA) is a protein made by the prostate gland and found in the blood. PSA blood levels may be higher than normal in men who have prostate cancer, benign prostatic hyperplasia (BPH), or infection or inflammation of the prostate gland, and are often used to monitor patients who have been treated for prostate cancer to see if their cancer has recurred.
  ng/ml | 0.32 [0.1 to 1.96] | 0.40 [0.1 to 1.93] | 0.32 [0.1 to 1.93] | 0.35 [0.1 to 1.96]
Pre-RT Entry PSA [Count of Participants; unit: Participants]
  >= 0.1 and <= 0.2 ng/ml | 155 | 126 | 154 | 435
  > 0.2 and <= 0.5 ng/ml | 247 | 256 | 247 | 750
  > 0.5 and <= 1.0 ng/ml | 105 | 130 | 114 | 349
  > 1.0 and < 2.0 ng/ml | 57 | 66 | 59 | 182

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Free From Progression (FFP) at 5 Years
Description: Progression is defined as the first occurrence of the following events: biochemical failure by the Phoenix definition (prostate-specific antigen [PSA] ≥ 2 ng/ml over the nadir PSA), clinical failure (local, regional or distant), or death from any cause. The initiation of second salvage therapy before progression was a protocol violation and resulted in censoring. Progression time is defined as time from randomization to the date of progression, second salvage therapy (censored), or last known follow-up (censored). Freedom from progression rates are estimated using the Kaplan-Meier method. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but results were reported early. See Limitations and Caveats section.
Time Frame: From randomization to five years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- PBRT Alone: (Arm 1) Prostate bed radiotherapy (PBRT) begins within 6 weeks (+/- 2 weeks) after registration.
- PBRT + STAD: (Arm 2) Prostate bed radiotherapy (PBRT) and short term androgen deprivation therapy (STAD) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STAD starts first, 2 months (+/- 2 weeks) before radiotherapy (RT), and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
- PLNRT + PBRT + STAD: (Arm 3) Pelvic lymph node radiotherapy (PLNRT), prostate bed radiotherapy (PBRT), and short term androgen deprivation therapy (STAD) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STAD starts first, 2 months (+/- 2 weeks) before RT, and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 70.3 [66.2 to 74.3] | 81.3 [77.9 to 84.6] | 87.4 [84.6 to 90.3]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Alternative hypotheses: 10% improvement in 5-year FFP in Arm 2 and 20% improvement in Arm 3, both relative to Arm 1, which has an assumed 5-year FFP of 70%. Sample size of 1587 (529/arm) with overall one-sided 0.025 alpha provides 90% power. Interim analyses (reported here) tested at one-sided significance level of 0.001. P<0.001 indicates comparison crossed interim efficacy boundary. See Limitations and Caveats section; Test type: Superiority; p < 0.001, Z test — One-sided significance level = 0.001
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.003, Z-test
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.001, Z-test

2. Secondary Outcome: Percentage of Participants With Secondary Biochemical Failure (Alternative Biochemical Failure)
Description: Secondary biochemical (failure) is defined as either of two occurrences: 1. For detectable post-baseline PSA values (≥ 0.1), the first occurrence of a PSA value that is both ≥ 0.4 and a second rise above nadir; 2.The start of second salvage therapy. Failure time is defined as time from randomization to the date of failure, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but results were reported early. See Limitations and Caveats section.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 35.7 [31.6 to 39.9] | 22.3 [18.8 to 26.0] | 14.5 [11.6 to 17.7]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.57, 97.5% CI 2-sided [0.45 to 0.72] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.67, 97.5% CI 2-sided [0.51 to 0.89] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.39, 97.5% CI 2-sided [0.30 to 0.51] — Reference level = PBRT Alone

3. Secondary Outcome: Percentage of Participants Free From Hormone-refractory Disease (Castrate-resistant Disease)
Description: Hormone-refractory disease (failure) is defined as three rises in PSA after the start of second salvage androgen deprivation therapy. Failure time is defined as time from randomization to the date of failure, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but the data monitoring committee decided to release results after the third interim analysis.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 2.9 [1.7 to 4.7] | 2.4 [1.3 to 4.1] | 1.2 [0.5 to 2.5]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p = 0.137, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.73, 97.5% CI 2-sided [0.39 to 1.39] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.007, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.39, 97.5% CI 2-sided [0.16 to 0.95] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.29, 97.5% CI 2-sided [0.12 to 0.68] — Reference level = PBRT Alone

4. Secondary Outcome: Percentage of Participants With Local Failure
Description: Local failure is defined as first occurrence of local clinical progression. Failure time is defined as time from randomization to the date of failure, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but the data monitoring committee decided to release results after the third interim analysis.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 3.1 [1.8 to 4.9] | 1.2 [0.5 to 2.4] | 0.4 [0.1 to 1.3]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p = 0.010, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.37, 97.5% CI 2-sided [0.14 to 1.01] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.177, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.56, 97.5% CI 2-sided [0.14 to 2.30] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.21, 97.5% CI 2-sided [0.06 to 0.71] — Reference level = PBRT Alone

5. Secondary Outcome: Percentage of Participants With Distant Metastasis
Description: Distant metastasis (failure) is defined as the occurrence of distant metastasis determined by imaging. Failure time is defined as time from randomization to the date of failure, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but the data monitoring committee decided to release results after the third interim analysis.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 8.3 [6.1 to 11.0] | 5.9 [4.1 to 8.2] | 4.7 [3.1 to 6.8]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p = 0.105, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.78, 97.5% CI 2-sided [0.49 to 1.22] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.022, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.62, 97.5% CI 2-sided [0.36 to 1.06] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p < 0.001, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.48, 97.5% CI 2-sided [0.29 to 0.81] — Reference level = PBRT Alone

6. Secondary Outcome: Percentage of Participants Who Died Due to Prostate Cancer (Cause-specific Mortality)
Description: Cause-specific mortality (failure) is defined as death due to prostate cancer or complications of protocol treatment (centrally reviewed), or death following disease progression (clinical or biochemical) in the absence of or after the initiation of any salvage therapy. [Biochemical progression is indicated by any rise in PSA.] Failure time is defined as time from randomization to the date of failure, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but the data monitoring committee decided to release results after the third interim analysis.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 2.7 [1.5 to 4.4] | 1.1 [0.4 to 2.3] | 0.8 [0.3 to 1.9]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p = 0.137, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.71, 97.5% CI 2-sided [0.35 to 1.43] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.141, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.68, 97.5% CI 2-sided [0.30 to 1.54] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.014, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.47, 97.5% CI 2-sided [0.21 to 1.03] — Reference level = PBRT Alone

7. Secondary Outcome: Percentage of Participants Alive (Overall Mortality)
Description: Survival time is defined as time from randomization to the date of death from any cause or last known follow-up (censored). Survival rates are estimated by the Kaplan-Meier method. Pairwise comparisons of the overall distributions of failure times are reported in statistical analysis section, with five-year rates reported here. The study was designed for the final analysis to occur after all participants had been on study for at least 5 years, but the data monitoring committee decided to release results after the third interim analysis.
Time Frame: From randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants | 93.9 [91.8 to 96.0] | 96.1 [94.4 to 97.8] | 95.7 [94.0 to 97.4]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Test type: Superiority; p = 0.235, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.86, 97.5% CI 2-sided [0.54 to 1.38] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.481, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.99, 97.5% CI 2-sided [0.61 to 1.60] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PLNRT + PBRT + STAD; Test type: Superiority; p = 0.213, Log Rank — One-sided significance level = 0.0125; Hazard Ratio (HR) = 0.85, 97.5% CI 2-sided [0.53 to 1.35] — Reference level = PBRT Alone

8. Secondary Outcome: Percentage of Participants Experiencing Grade 2+ and 3+ Adverse Events ≤ 90 Days of the Completion of Radiotherapy (RT)
Description: Common Terminology Criteria for Adverse Events (version 3.0) grades adverse event severity from 1=mild to 5=death. Summary data is provided in this outcome measure; see Adverse Events Module for specific adverse event data. Pairwise comparisons of Arm 2 vs Arm 1 and Arm 3 vs. Arm 2 are reported in the statistical analysis.
Time Frame: From randomization to 90 days after completion of radiotherapy (approximately 7-8 weeks).
Population: Eligible participants
Measure: Number; unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants
  Grade 2+ | 18.8 | 36.3 | 43.6
  Grade 3+ | 4.4 | 8.7 | 12.2
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Acute grade 2+ acute adverse events; Test type: Superiority; p < 0.001, Regression, Logistic — One-sided significance level = 0.025; Model was adjusted for entry PSA level, pathology, seminal vesicle involvement, Gleason score, race, and age; Odds Ratio (OR) = 2.47, 97.5% CI 2-sided [1.81 to 3.37] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Acute grade 2+ acute adverse events; Test type: Superiority; p = 0.007, Regression, Logistic — One-sided significance level = 0.025; Model was adjusted for entry PSA level, pathology, seminal vesicle involvement, Gleason score, race, and age; Odds Ratio (OR) = 1.35, 97.5% CI 2-sided [1.03 to 1.77] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PBRT + STAD; Acute grade 3+ acute adverse events; Test type: Superiority; p = 0.002, Regression, Logistic — One-sided significance level = 0.025; Univariate model was used due to the low number of events; Odds Ratio (OR) = 2.04, 97.5% CI 2-sided [1.16 to 3.60] — Reference level = PBRT Alone
Statistical Analysis 4: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Acute grade 3+ adverse events; Test type: Superiority; p = 0.025, Regression, Logistic — One-sided significance level = 0.025; Univariate model was used due to the low number of events; Odds Ratio (OR) = 1.47, 95% CI 2-sided [0.975 to 2.27] — Reference level = PBRT + STAD

9. Secondary Outcome: Percentage of Participants Experiencing Late Grade 2+ and 3+ Adverse Events > 90 Days From the Completion of Radiotherapy (RT)
Description: Common Terminology Criteria for Adverse Events (version 3.0) grades adverse event severity from 1=mild to 5=death. Late adverse events (AE) are defined as occurring > 90 days from the completion of RT. Failure time is defined as time from randomization to the date of first late grade 2 or grade 3 adverse event, death (competing risk), or last known follow-up (censored). Failure rates for data summary are estimated using the cumulative incidence method, with 5-year rates provided here. Pairwise comparisons of the distributions of failure times between Arm 2 and Arm 1 and between Arm 3 and Arm 2, reported in the statistical analysis section, use cause-specific hazard rates for which deaths are censored.
Time Frame: AE: from 91 days after completion of RT (approximately 7-8 weeks) to last follow-up. Vital status: from randomization to last follow-up. Maximum follow-up at time of analysis was 10.5 years.
Population: Eligible participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | PBRT Alone | PBRT + STAD | PLNRT + PBRT + STAD
Number analyzed (Participants) | 564 | 578 | 574
percentage of participants
  Grade 2+ | 52.8 [48.4 to 57.0] | 54.8 [50.4 to 58.9] | 58.6 [54.3 to 62.6]
  Grade 3+ | 10.3 [7.8 to 13.2] | 11.4 [8.9 to 14.3] | 14.4 [11.6 to 17.5]
Statistical Analysis 1: Comparison: PBRT Alone vs PBRT + STAD; Late grade 2+ adverse events; Test type: Superiority; p = 0.268, Log Rank — One-sided significance level = 0.025; Hazard Ratio (HR) = 1.05, 97.5% CI 2-sided [0.88 to 1.26] — Reference level = PBRT Alone
Statistical Analysis 2: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Late grade 2+ adverse events; Test type: Superiority; p = 0.101, Log Rank — One-sided significance level = 0.025; Hazard Ratio (HR) = 1.10, 97.5% CI 2-sided [0.93 to 1.32] — Reference level = PBRT + STAD
Statistical Analysis 3: Comparison: PBRT Alone vs PBRT + STAD; Late grade 3+ adverse events; Test type: Superiority; p = 0.119, Log Rank — One-sided significance level = 0.025; Hazard Ratio (HR) = 1.22, 97.5% CI 2-sided [0.83 to 1.80] — Reference level = PBRT Alone
Statistical Analysis 4: Comparison: PBRT + STAD vs PLNRT + PBRT + STAD; Late grade 3+ adverse events; Test type: Superiority; p = 0.170, Log Rank — One-sided significance level = 0.025; Hazard Ratio (HR) = 1.16, 97.5% CI 2-sided [0.82 to 1.65] — Reference level = PBRT + STAD

10. Secondary Outcome: Comparison of Disease-specific Health Related Quality of Life (HRQOL) Change by the Expanded Prostate Cancer Index Composite (EPIC), Hopkins Verbal Learning Test Revised (HVLT-R), Trail Making Test A & B, and Controlled Oral Word Association Test (COWAT)
Time Frame: From the 6th week of radiation therapy to 5 years post radiation therapy.
Reporting Status: Not Posted, anticipated posting 2026-01

11. Secondary Outcome: Assessment of Mood and Depression Change Using QOL Measured by the Hopkins Symptom Checklist (HSCL-25)
Time Frame: From the 6th week of radiation therapy to 5 years post radiation therapy.
Reporting Status: Not Posted, anticipated posting 2026-01

12. Secondary Outcome: Assessment and Comparison of Quality Adjusted Life Year (QALY) and Quality Adjusted FFP Year (QAFFPY)
Time Frame: From the 6th week of radiation therapy to 5 years post radiation therapy.
Reporting Status: Not Posted, anticipated posting 2026-01

13. Secondary Outcome: Evaluation and Comparison of the Cost-utility Using EuroQoL - 5 Dimensions (EQ-5D)
Time Frame: From the 6th week of radiation therapy to 5 years post radiation therapy.
Reporting Status: Not Posted, anticipated posting 2026-01

14. Secondary Outcome: Prognostic Value of Genomic and Proteomic Markers for the Primary and Secondary Clinical Endpoints
Time Frame: Date of randomization to timepoint of the respective primary or secondary endpoint.
Reporting Status: Not Posted, anticipated posting 2026-01

15. Secondary Outcome: Assessment of the Relationship(s) Between the American Urological Association Symptom Index (AUA SI) and Urinary Morbidity (Adverse Event Terms: Urinary Frequency/Urgency) Using the CTCAE v. 3.0 Grading System
Time Frame: From the 6th week of radiation therapy to 5 years post radiation therapy.
Reporting Status: Not Posted, anticipated posting 2026-01

ADVERSE EVENTS:
Time Frame: Weekly during radiotherapy, at 3, 6, and 12 months after end of radiotherapy, every 6 months from end of treatment for 6 years, then annually until study completion. Maximum follow-up at time of reporting was 10.5 years.
Description: Eligible participants who started study treatment and have adverse event data.
Groups:
- PBRT + STADT: Prostate bed radiotherapy (PBRT) and short term androgen deprivation therapy (STADT) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STADT starts first, 2 months (+/- 2 weeks) before radiotherapy (RT), and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
- PLNRT + PBRT + STADT: Pelvic lymph node radiotherapy (PLNRT), prostate bed radiotherapy (PBRT), and short term androgen deprivation therapy (STADT) consisting of antiandrogen (AA) and luteinizing hormone-releasing hormone (LHRH) agonist therapy begins within 6 weeks (+/- 2 weeks) after registration. STADT starts first, 2 months (+/- 2 weeks) before RT, and lasts for 4-6 months. LHRH can last 4-6 months. AA starts at the same time as LHRH (or up to 2 weeks prior ), lasts approximately 4 months, and should end on the last day of RT (+/- 2 weeks).
Arm/Group | PBRT Alone | PBRT + STADT | PLNRT + PBRT + STADT
All-Cause Mortality (participants affected / at risk) | 48/547 | 43/563 | 43/563
Serious Adverse Events (participants affected / at risk) | 18/547 | 29/563 | 23/563
Other Adverse Events (participants affected / at risk) | 433/547 | 492/563 | 509/563
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBRT Alone (N=547) | PBRT + STADT (N=563) | PLNRT + PBRT + STADT (N=563)
Blood disorder (Blood and lymphatic system disorders) | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 1 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1 | 0
Myocardial ischemia (Cardiac disorders) | 1 | 2 | 0
Pericarditis (Cardiac disorders) | 0 | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Eye disorder (Eye disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Anal pain (Gastrointestinal disorders) | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2 | 1
Esophageal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Esophageal mucositis (Gastrointestinal disorders) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1 | 0
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Fatigue (General disorders) | 2 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Bladder infection [with unknown ANC] (Infections and infestations) | 1 | 1 | 0
Bone infection [with unknown ANC] (Infections and infestations) | 1 | 0 | 0
Infection [other] (Infections and infestations) | 0 | 1 | 1
Sepsis [with unknown ANC] (Infections and infestations) | 0 | 0 | 1
Urinary tract infection [with unknown ANC] (Infections and infestations) | 3 | 0 | 0
Intraoperative complications (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Ischemia cerebrovascular (Nervous system disorders) | 1 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 1
Bladder hemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Bladder obstruction (Renal and urinary disorders) | 1 | 0 | 0
Bladder stenosis (Renal and urinary disorders) | 1 | 0 | 0
Cystitis (Renal and urinary disorders) | 2 | 4 | 3
Hemorrhage urinary tract (Renal and urinary disorders) | 0 | 1 | 0
Renal hemorrhage (Renal and urinary disorders) | 1 | 0 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1 | 0
Urethral obstruction (Renal and urinary disorders) | 0 | 2 | 0
Urethral stricture (Renal and urinary disorders) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 3 | 2
Urinary incontinence (Renal and urinary disorders) | 4 | 1 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1 | 1
Urogenital disorder (Renal and urinary disorders) | 5 | 2 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Skin disorder (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0
Lymphocele (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PBRT Alone (N=547) | PBRT + STADT (N=563) | PLNRT + PBRT + STADT (N=563)
Hemoglobin decreased (Blood and lymphatic system disorders) | 32 | 73 | 80
Constipation (Gastrointestinal disorders) | 54 | 53 | 59
Diarrhea (Gastrointestinal disorders) | 110 | 127 | 219
Gastrointestinal disorder (Gastrointestinal disorders) | 36 | 36 | 33
Hemorrhoids (Gastrointestinal disorders) | 26 | 29 | 33
Proctitis (Gastrointestinal disorders) | 62 | 55 | 66
Rectal hemorrhage (Gastrointestinal disorders) | 43 | 50 | 48
Fatigue (General disorders) | 148 | 211 | 217
Pain [other] (General disorders) | 30 | 31 | 43
Alanine aminotransferase increased (Investigations) | 8 | 35 | 23
Aspartate aminotransferase increased (Investigations) | 11 | 35 | 20
Leukopenia (Investigations) | 32 | 29 | 40
Lymphopenia (Investigations) | 28 | 26 | 50
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 35 | 26
Libido decreased (Psychiatric disorders) | 35 | 67 | 83
Cystitis (Renal and urinary disorders) | 69 | 72 | 71
Hemorrhage urinary tract (Renal and urinary disorders) | 36 | 29 | 36
Urinary frequency (Renal and urinary disorders) | 281 | 333 | 348
Urinary incontinence (Renal and urinary disorders) | 237 | 215 | 239
Urinary retention (Renal and urinary disorders) | 69 | 69 | 78
Urogenital disorder (Renal and urinary disorders) | 77 | 64 | 80
Erectile dysfunction (Reproductive system and breast disorders) | 155 | 185 | 202
Hot flashes (Vascular disorders) | 36 | 327 | 325

LIMITATIONS AND CAVEATS:
Three interim analyses were planned when there were 397, 794, and 1191 eligible patients with five years of potential follow-up from the randomization date. Due to findings from the third interim analysis, the data monitoring committee recommended that study results be reported early for all arms, while recognizing that the originally planned full analysis will provide additional insight for the Arm 3 vs. Arm 2 comparison.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI's are required to abide by the sponsor's publication guidelines which require review by coauthors and subsequent review and approval by the sponsor.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT00567580/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-01): https://cdn.clinicaltrials.gov/large-docs/80/NCT00567580/ICF_001.pdf